CLINICAL TRIAL: NCT02865980
Title: Effect of Washing With Clove Extract on Inflammation and Infection Place Logging Shaldon Needle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali bazzi, Mashhad Faculty of Nursing and Midwifery, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 95150200
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Renal Failure
Keywords: inflammation, infection
MeSH Terms: conditions — Renal Insufficiency; Inflammation; Infections | interventions — Phosphatidylinositol 3-Kinases; Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- inflammation (Experimental): The effect of washing with betadine and clove extract on incidence of inflammation place logging shaldon catheter in the hemodialysis patients
  Interventions: Other: clove extract; Other: Betadine
- infection (Experimental): The effect of washing with betadine and clove extract on incidence of infection place logging shaldon catheter in the hemodialysis patients
  Interventions: Other: clove extract; Other: Betadine

INTERVENTIONS:
Other: clove extract — in intervention group, first will be washed the Catheter with Betadine after 2 minutes will be used of the clove extract with 2 ml of scrub for 15 seconds. The incidence of inflammation of vascular access will be assessed in patients on hemodialysis for each patient before starting the process over a period of 2 weeks is equivalent to 6 sessions of hemodialysis.
Other: Betadine — in control group, will be washed the Catheter with Betadine

SUMMARY:
This randomized clinical trial will conducted involving 60 patients under hemodialysis and hospitalized to Imam Reza and Montasareyeh hospitals of Mashhad in 2016. Patients were assigned to experimental and control groups of 30 people, randomly (double block). In the both intervention and control group, first will be washed the Catheter with Betadine, but in intervention group, after 2 minutes will be used of the clove extract with 2 ml of scrub for 15 seconds. The incidence and severity of inflammation as well as infection of vascular access will be assessed in patients on hemodialysis for each patient before starting the process over a period of 2 weeks is equivalent to 6 sessions of hemodialysis.

DETAILED DESCRIPTION:
This study is a randomized clinical trial that will conducted on 60 patients under hemodialysis and hospitalized to Imam Reza and Montasareyeh hospitals of Mashhad in 2016. Patients were assigned to experimental and control groups of 30 people, randomly (double block).

In the both intervention and control group, first will be washed the shaldon catheter with Betadine, but in intervention group, after 2 minutes will be used of the clove extract with 2 ml of scrub for 15 seconds. The incidence and severity of inflammation as well as infection of vascular access will be assessed in patients on hemodialysis for each patient before starting the process over a period of 2 weeks is equivalent to 6 sessions of hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18-80

Exclusion Criteria:

* lack of cooperation patient to participate in the post test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
inflammation severity questionnaire | 6 weeks
  effects of washing with clove extract on inflammation place logging shaldon needles in the hemodialysis patients that will be measured with inflammation severity questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Bazzi, MSc, Principal Investigator — Mashhad Faculty Nursing and Midwifery
Locations (1):
- Mashhad Faculty of Nursing and Midwifery, Mashhad, Khorasan Razavi, Iran

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chaudhari LK, Jawale BA, Sharma S, Sharma H, Kumar CD, Kulkarni PA. Antimicrobial activity of commercially available essential oils against Streptococcus mutans. J Contemp Dent Pract. 2012 Jan 1;13(1):71-4. doi: 10.5005/jp-journals-10024-1098. PMID 22430697
- See also: abstract article — http://ncbi.nlm.nih.gov/pubmed/22430697